CLINICAL TRIAL: NCT00786825
Title: Measurement of Glucose/Glycogen Metabolism in Humans Using Magnetic Resonance at 4 or 7 Tesla
Acronym: Glycogen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9412M09040
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Hypoglycemia unawareness
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Somatostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- somatostatin (Experimental): Type 1 diabetes and Hypoglycemia unawareness
  Interventions: Drug: somatostatin
- 2 (No Intervention): Healthy control subjects

INTERVENTIONS:
Drug: somatostatin — Somatostatin may be used to suppress endogenous insulin secretion
  Arms: somatostatin

SUMMARY:
The long-range goal of this project is to determine the effects of diabetes and the hypoglycemic consequences of intensive therapy on in vivo brain glucose metabolism in humans. We will measure brain glycogen turnover and content in normal controls and subjects with diabetes under conditions of modest hyper-and hypoglycemia.

DETAILED DESCRIPTION:
On the morning before the study subjects will report to the Clinical Research Center and will be asked to stay at the Clinical Research Center for up to 72 hours. You will be asked not to eat anything after midnight. Small plastic catheters will be placed in two veins in subjects arms for infusion of glucose and for measuring blood glucose levels every 15-30 minutes. While subjects are in the study they will continuously receive a small dose of glucose enriched with 13C label either through the catheter or by drinking a small amount of a sugar water solution every 15-60 minutes. Subjects will be asked to transfer to the Center for Magnetic Resonance Research every 6-8 hours (except at night) where they will be asked each time to conduct an MRI scan as follows: Subjects will be placed on the patient bed in the magnet room for one-to-two hours. A nurse will stay with the subject at all times during this study. During some of the scans subjects may be asked to perform a visual task such as watching a changing checkerboard pattern through a mirror placed in front of their eyes. After each scan subjects will receive a low carbohydrate meal for weight-maintenance.

Subjects may be asked to receive an infusion of glucose and/or insulin one-to-three times before and/or after the infusion of 13C-enriched glucose starts. During these infusions the subject's blood sugar will be maintained either higher or lower than normal levels for up to 3 hours. This will be done to assess the effect of hyper- or hypoglycemia on brain glycogen metabolism.

Subjects may also be asked several days prior to the study to report to the Clinical Research Center for a "mock" study to see if they are comfortable with the MRI scan and/or to test their body's response to either protocol (as described above, but carried out at the Clinical Research Center). If subjects would like to try the MRI procedure in advance, this test will not exceed 2 hours. If we need to test the subject's response to the infusion, this "pre-test" will involve only drawing blood and administering glucose and will be performed as described for either protocol above, but will last not more than 4 hours.

Magnetic resonance measurements will be performed in the magnet and are very similar to magnetic resonance imaging exams (MRI). Subjects will always have the possibility to signal when they feel claustrophobic and wish to be removed from the magnet. The magnetic resonance measurements will be associated with a regular clunking noise that subjects may initially find unpleasant. For their comfort they will be offered to wear ear plugs. During the measurements in the magnet subjects will be asked to lie still for most of the time.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Healthy control
* Must be able to provide informed consent
* Type 1 diabetes with hypoglycemia unawareness with hemoglobin A1c < 7.5%
* Poorly controlled diabetics with hemoglobin A1c > 7.5%
* Subjects with hypoglycemia unawareness must report an inability to recognize at least some blood glucose values <58 mg/dL during the 3 months prior to the study.

Exclusion Criteria:

* Over 300 pounds
* Claustrophobic
* History of ischemic heart disease, arrhythmia, of seizure disorder
* Pregnant
* On medications known to alter blood flow or carbohydrate metabolism
* Have internally located pieces of metal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Seaquist, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Seaquist ER, Moheet A, Kumar A, Deelchand DK, Terpstra M, Kubisiak K, Eberly LE, Henry PG, Joers JM, Oz G. Hypothalamic Glucose Transport in Humans During Experimentally Induced Hypoglycemia-Associated Autonomic Failure. J Clin Endocrinol Metab. 2017 Sep 1;102(9):3571-3580. doi: 10.1210/jc.2017-00477. PMID 28911152

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls: Healthy control subjects
Period: Overall Study
Arm/Group | Somatostatin | Healthy Controls
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Somatostatin | Healthy Controls | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (4) | 57 (3) | 57 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Brain Glycogen Turnover Rate
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Somatostatin | Healthy Controls
Number analyzed (Participants) | 5 | 5
mg/kg/min | 0.31 (0.23) | 0.28 (0.06)

ADVERSE EVENTS:
Time Frame: Course of study, 1 month
Arm/Group | Somatostatin | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2014-04-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT00786825/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2011-09-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT00786825/Prot_SAP_001.pdf